CLINICAL TRIAL: NCT00490750
Title: Randomized Prospective Trial of Laparoscopic Heller Myotomy and Partial Fundoplication for the Treatment of Idiopathic Esophageal Achalasia
Brief Title: Laparoscopic Dor Versus Toupet Fundoplication for the Treatment of Idiopathic Esophageal Achalasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: L. Michael Brunt (Other)
Collaborators: University of Washington (Other); Northwestern University (Other); University of Oregon (Other); Duke University (Other)
Responsible Party: Sponsor-Investigator, L. Michael Brunt, Professor of Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 03-0241
Record Dates: First submitted 2007-06-21; First posted 2007-06-25 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Esophageal Achalasia
Keywords: Heller Dor; Heller Toupet; Myotomy
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic Dor fundoplication (Active Comparator): Heller myotomy followed by Dor fundoplication
  Interventions: Procedure: Dor fundoplication
- Laparoscopic Toupet fundoplication (Active Comparator): Heller myotomy followed by Toupet fundoplication
  Interventions: Procedure: Toupet fundoplication

INTERVENTIONS:
Procedure: Dor fundoplication — Subjects are randomized to undergo Heller myotomy followed by Laparoscopic Dor fundoplication
  Arms: Laparoscopic Dor fundoplication
Procedure: Toupet fundoplication — Subjects are randomized to undergo Heller myotomy followed by Laparoscopic Toupet fundoplication
  Arms: Laparoscopic Toupet fundoplication

SUMMARY:
The primary aim of this study is to test the hypothesis that Heller myotomy and Toupet fundoplication result in a lower rate of reflux symptoms and positive 24-hour pH testing when compared to Heller myotomy and Dor fundoplication.

DETAILED DESCRIPTION:
Idiopathic achalasia is an uncommon motor disorder of the esophagus which occasionally requires surgical intervention. Although there are several controversial aspects of therapy for achalasia, laparoscopic myotomy is emerging as the procedure of choice. Several studies report having good to excellent outcomes following a laparoscopic procedure in approximately 90% of patients. However, a main deterrent to long-term success is the development of gastroesophageal reflux disease (GERD) despite the use of an antireflux procedure. For this reason, most surgeons add a partial fundoplication to the myotomy. The gastric fundus can either be wrapped anterior to the esophagus (Dor fundoplication), or posterior to the esophagus (Toupet fundoplication). Currently, the type of fundoplication is determined by surgeon's choice. There exists no systematic comparison of the two procedures. This multicenter, randomized study aims to evaluate patient outcomes following myotomy and Dor versus Toupet fundoplication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Achalasia

Exclusion Criteria:

* Prior heller myotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Primary outcomes are 24 hour pH testing results | pH testing at 6-12 months after surgical treatment

SECONDARY OUTCOMES:
Symptomatic response measured by detailed patient questionnaire and results of barium swallow radiographs | 6-12 months after surgical intervention

CONTACTS AND LOCATIONS:
Overall Officials: L. Michael Brunt, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States